CLINICAL TRIAL: NCT02184390
Title: Parenting Your Young Child With Autism: A Web-Based Tutorial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Psychological Consultation (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kenneth A. Kobak, Ph.D., Principal Investigator, Center for Psychological Consultation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R44MH086936 (NIH); 5R44MH086936 (NIH)
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Autistic Disorder
Keywords: Internet; Education
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tutorial (Experimental): Parents who receive access to the tutorial immediately
  Interventions: Other: On LIne Parent Training Tutorial
- wait list control (No Intervention): Parents who are assessed at the same time points as the intervention arm, but do no receive access to the tutorial

INTERVENTIONS:
Other: On LIne Parent Training Tutorial — Interactive on line tutorial for parenting skills for autism
  Arms: tutorial

SUMMARY:
This study will evaluate the efficacy and user satisfaction with a web-based interactive tutorial for caregivers of young children with autism designed to a) teach parents how to promote their child's development in the core deficit areas, b) help parents understand and improve challenging behaviors their child may demonstrate, and c) reduce caregiver stress through more effective interactions. It emphasizes everyday situations as opportunities for learning, including common home routines and contains videotaped illustrations of parents using the techniques taught in the home environment.

DETAILED DESCRIPTION:
Autism is a neurodevelopmental disorder characterized by core deficits in social reciprocity, verbal and nonverbal communication, and behavior. Early detection and intervention has been shown to improve these core deficits, resulting in better long-term outcomes in language functioning, cognitive/developmental skills, and social and adaptive behavior. Despite the demonstrated benefits of effective intervention, few children receive these specialized services, due in part to critical resource barriers, such as the shortage of specialists trained to deliver them. The broad, long-term objective of this project is to improve outcomes for children with autism and their families by empowering caregivers with the knowledge and skills needed to effectively intervene directly with their children as part of their daily interactions and routines. By targeting those with the most invested in the child's success and the longest lasting influence on a child's long-term growth and development, we can help parents in several ways: a) teach parents how to promote their child's development in the core deficit areas seen in young children with autism spectrum disorders: social interaction, communication, play, and imitation; b) help parents understand and improve challenging behaviors their child may demonstrate, and c) reduce caregiver stress through more effective interactions.

To make this training widely accessible to parents of children with autism, we will deliver this training through a web-based, multi-media, interactive tutorial. The tutorial will use principles of instructional design to more effectively deliver the material and utilize high levels of interactivity afforded by the web-based platform to maximize learning. The tutorial teaches skills to improve their child's behavior and communication within the framework of everyday routines and activities, utilizing interactive exercises and a comprehensive set of videos of real parents implementing these strategies with their children within the context of everyday situations.

The specific aims of the proposed Phase II study are:

Aim 1. To evaluate parents' satisfaction and acceptance of the tutorial program Aim 2. To demonstrate the tutorial increases parental knowledge of the principles and techniques for improving effective parenting of children with Autism Spectrum Disorder.

Aim 3. To demonstrate behavioral improvements in actual parenting skills during the daily interactions with their child based on the knowledge gained.

Aim 4. To demonstrate that the improved parenting skills result in social, communication, and behavioral improvements in the children of parents who complete the tutorial.

Aim 5. To demonstrate that improving parenting skills through the use of this web-based tutorial program reduces caregiver stress and depression.

ELIGIBILITY:
Inclusion Criteria:

* parents or caregivers of children with ASD between the ages of 18 months and 6 years with an autism spectrum disorder

Exclusion Criteria:

* Ability to read and understand English

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2013-05; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
System Usability Scale | 8 weeks
  User satisfaction with the technical aspects of the Enhancing Interactions tutorial will be assessed using the ratings on the System Usability Scale (SUS). The SUS is a reliable, well-validated 10-item scale 1,49 designed to evaluate the usability and user satisfaction with web-based applications and other technologies. It yields quantitative feedback on a 0-100 scale regarding the effectiveness, efficiency, and satisfaction of users while interacting with engineered systems.

SECONDARY OUTCOMES:
Autism Knowledge Test | 8 weeks
  Gains in parents' knowledge regarding of the principles and techniques for more effective parenting of children will be demonstrated using a pre and post test of 24-items developed by the content experts (Drs. Stone and Warren, and Lisa Wallace) that covers the core concepts of the tutorials. The test items were piloted in parents who (a) had received face-to-face training during Enhancing Interactions seminars and (b) other parents prior to being trained. Items were selected based on their psychometric properties and sensitivity to discriminate between parents who had and had not been exposed to the Enhancing Interactions training.

OTHER OUTCOMES:
The Parent Interview for Autism-Clinical Version | 8 weeks
Parenting Efficacy Scale | 8 weeks
Parenting Stress Index | 8 weeks
Child and Parent Behavior Form | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Psychological Consulation, Madison, Wisconsin, United States

REFERENCES:
- [Background] Kobak KA, Stone WL, Wallace E, Warren Z, Swanson A, Robson K. A web-based tutorial for parents of young children with autism: results from a pilot study. Telemed J E Health. 2011 Dec;17(10):804-8. doi: 10.1089/tmj.2011.0060. Epub 2011 Oct 19. PMID 22011005